CLINICAL TRIAL: NCT04993053
Title: Use of Cemented TFNA Nail Augmentation in the Treatment of Trochanterian Rock Fractures in Patients Over 65 Years of Age
Brief Title: Use of Cemented TFNA Nail Augmentation in the Treatment of Trochanterian Rock Fractures
Acronym: TFNA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: TFNA - 29BRC21.0076
Record Dates: First submitted 2021-07-06; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: the Cement Augmented Screws of TFNA Nails
Keywords: TFNA; Hip fracture; Augmentation; Cement; Cut-out
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intramedullary nailing is the standard treatment of trochanteric fractures. Mechanical failure such as cut-out and cut-through are associated with high rates of revision surgery, functional impairment and mortality. Augmentation of the implant have shown encouraging results in reducing the number of mechanical failures. The aim of the study was to evaluate the rate of mechanical failure of the cement augmented screws of TFNA nails.

A descriptive, retrospective, multi-operator, single-centre study was performed at our level 1 trauma centre. Patients were included if they were > 65 years of age, presented with a trochanteric fracture treated with an augmented TFNA nail. The primary outcome was fixation failure rate (cut-out or cut-through) at 3 and 6 postoperative months. Secondary endpoints were intraoperative data, clinical scores, and radiographic analysis.

ELIGIBILITY:
Inclusion Criteria:

* > 65 years of age
* a trochanteric fracture that occurred through a low-energy mechanism
* an augmented TFNA nail

Exclusion Criteria:

* pathological fracture
* open fracture
* hips with pre-existing deformities other than osteoarthritis
* a history of hip surgery
* an insufficient quantity of injected cement (< 3 mL).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consisted of 61 patients. The analyses were therefore based on 45 patients (Table 1). The 38 women and 7 men had a mean age of 82.84 years (65-102, 9.50) and most had sustained AO/OTA 31-A1.2 fractures.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Fixation failure rate (cut-out or cut-through) | change at 3 and 6 postoperative months
  On X rays

SECONDARY OUTCOMES:
Visual Analogue Scale score | at 3 and 6 postoperative months
  the minimum is 0 and maximum 10, higher scores mean a worse outcome.
analysis evaluating quality of reduction | once
  On X rays
Augmentation volume | once
length of surgery | at 3 and 6 postoperative months
radiation exposure | once
duration of hospitalisation | once
Intraoperative adverse events | once
EuroQoL 5-Dimensions score | change at 3 and 6 postoperative months
  the minimum is 5 and maximum 15, higher scores mean a worse outcome.
Parker Mobility Score | at 3 and 6 postoperative months
  the minimum is 0 and maximum 9, higher scores mean a better outcome.
Harris Hip Score | at 3 and 6 postoperative months
  the minimum is 0 and maximum 100, higher scores mean a betteroutcome.
the tip-apex distance | once
  On X rays
TFNA screw position | once
  On X rays
distribution of cement on either side of the cervicocephalic screw | once
  On X rays
postoperative complications | at 3 and 6 postoperative months
the need for revision surgery | at 3 and 6 postoperative months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending five years following the final study report completion.
Access Criteria: Data access request will be reviewed by the internal committee of Brest University Hospital. Requestor will be required to sign and complete a data access agreement.